CLINICAL TRIAL: NCT05922033
Title: Patient Versus Provider-led Titration of Insulin for Glycemic Control in Gestational Diabetes
Brief Title: Patient Versus Provider-led Titration of Insulin for Glycemic Control in Gestational Diabetes (EMPOWER)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kartik K Venkatesh, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023H0222
Record Dates: First submitted 2023-06-14; First posted 2023-06-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy in Diabetic; Pregnancy, High Risk
Keywords: Titration of insulin; Pregnancy; Glycemic control
MeSH Terms: conditions — Diabetes, Gestational; Pregnancy in Diabetics | interventions — Insulin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patient-led self-titration of insulin (Experimental): Individuals randomized to this arm will initiate night-time insulin of 10 units. The type of basal insulin will be left to the discretion of the provider with levemir or glargine preferred over NPH. On day 0 of initiation of insulin, the patient will initiate night-time (or prior to sleep if alternate sleep schedule) insulin of 10 units (glargine, detemir, or NPH). Patient will check their fasting blood glucose in the morning and record their values. If the value is below 70 they will decrease their insulin dosage that night by 2 units; if the value is above 95 they will increase their insulin dosage that night by 2 units; and if the value is between 70 and 95, they will maintain the same insulin dosage that night. The patients will continue this algorithm for the remainder of the pregnancy. If the patient does not have a fasting blood glucose, the patient will maintain the dose of basal insulin at the prior dose.
  Interventions: Drug: Patient-led Insulin (intervention group)
- Standard of care (Active Comparator): Individuals randomized to this arm will receive standard care and titration of insulin will be determined by the individual providers.
  Interventions: Drug: Provider-led Insulin (standard care)

INTERVENTIONS:
Drug: Patient-led Insulin (intervention group) — Individuals randomized to this arm will initiate night-time insulin of 10 units. The type of basal insulin will be left to the discretion of the provider with levemir or glargine preferred over NPH. On day 0 of initiation of insulin, the patient will initiate night-time (or prior to sleep if alternate sleep schedule) insulin of 10 units (glargine, detemir, or NPH). Patient will check their fasting blood glucose in the morning and record their values. If the value is below 70 they will decrease their insulin dosage that night by 2 units; if the value is above 95 they will increase their insulin dosage that night by 2 units; and if the value is between 70 and 95, they will maintain the same insulin dosage that night. The patients will continue this algorithm for the remainder of the pregnancy. If the patient does not have a fasting blood glucose, the patient will maintain the dose of basal insulin at the prior dose.
  Other Names: insulin
  Arms: Patient-led self-titration of insulin
Drug: Provider-led Insulin (standard care) — Individuals randomized to this arm will receive standard care and titration of insulin will be determined by the individual providers.
  Other Names: insulin
  Arms: Standard of care

SUMMARY:
We propose a pragmatic, unblinded, randomized controlled, single center trial of 56 pregnant individuals with Gestational diabetes mellitus (GDM). Our study proposes a pragmatic randomized control trial of patient led rapid titration of basal insulin compared to standard therapy. There is a planned subgroup analysis of patients with and without concomitant metformin usage. Patients will continue routine clinic visits. Patients who are initiated on basal insulin or started on night-time basal insulin within 7 days will be approached about the study. Patients who agree to be enrolled will sign informed consent.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is one of the most frequent medical complications of pregnancy and affects nearly 1 in 10 pregnant individuals. GDM is associated with an increased risk of adverse pregnancy outcomes for both the pregnant individual (cesarean delivery, preeclampsia) and infant (large for gestational age at birth, preterm birth <37 weeks, neonatal hypoglycemia, and hyperbilirubinemia). Improved glycemic control has been associated with reduction in the risks of these adverse pregnancy outcomes. Nearly 1 in 4 pregnant individuals with GDM will require medication to achieve glycemic control. The first-line therapy historically recommended for glycemic control is insulin and continues to be the primary recommendation of guidelines from the American College of Obstetrics and Gynecology (ACOG) and the American Diabetes Association (ADA). However current guidelines do not recommend a clear approach to insulin titration in GDM. This is an important limitation of current clinical practice. Individuals with GDM who are generally diagnosed between 24 to 28 weeks only have a short window of up to a few months to achieve glycemic control with pharmacotherapy to prevent adverse pregnancy outcomes. Traditionally, provider led titration of insulin has been the standard of care. Recommendations from outside of pregnancy and limited observational data from pregnancy have proposed patient-led self-titration of basal insulin have improved glycemic control compared to provider led titration.

We propose to conduct a pragmatic randomized controlled trial "EMPOWER: Patient versus provider-led titration of basal insulin for glycemic control in gestational diabetes" to compare pregnant individuals with GDM diagnosed >20 weeks gestation randomized to patient-led (intervention) versus provider-led insulin titration (standard of care).

OVERALL AIM: To conduct a pragmatic, non-blinded randomized controlled trial (pRCT) of patient-led insulin titration versus provider-led titration of basal insulin to improve glycemic control in the late third trimester in pregnancies complicated by gestational diabetes.

1.2 Specific Aims

PRIMARY AIM:

Compare glycemic control defined as the mean fasting glucose in the last week prior to term (36 weeks) between individuals randomized to patient-led (intervention) versus provider-led insulin titration (standard of care).

SECONDARY AIMS:

Secondary Aim 1: Compare the frequency of adverse pregnancy outcomes (cesarean delivery, preeclampsia, large for gestational age, and NICU admission) between individuals randomized to patient-led (intervention) versus provider-led insulin titration (standard of care).

Secondary Aim 2: Compare effect of concurrent metformin use on total daily insulin dose per kilogram at 36 weeks overall, and by patient-led (intervention) versus provider-led insulin titration.

Secondary Aim 3: Compare patient and provider satisfaction between patient-led (intervention) versus provider-led insulin titration.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant individuals with a diagnosis of Gestational diabetes mellitus (GDM) between 20 0/7 to 31 6/7 - 32 6/7 weeks and requiring initiation of basal insulin initiation as determined by provider
* Patients not on insulin or insulin initiation within 7 days of consent and randomization
* ≥ 18 years old with the ability to give informed consent
* Diagnosed with GDM during pregnancy by a one-hour 50-gram glucose challenge test ≥200 mg/dL at greater than 20 weeks of gestation or two elevated values on a 3-hour or a 100-gram glucose tolerance test at greater than 20 weeks of gestation.
* English or Spanish speaking
* Receiving prenatal care at OSU or an affiliated clinic where Electronic Health Records (EHR) can be accessed

Exclusion criteria:

* Type 1 or 2 diabetes
* Insulin allergy
* Not English or Spanish speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is restricted to pregnant individuals.
Enrollment: 56 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Fasting glycemic control | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  Continuous measure of mean fasting glucose during the 36th week of pregnancy. Patients with have the mean fasting glucose value during the 36th week of pregnancy. We will use this goal given that inadequate glycemic control may be delivered as soon as the early term period (37-39 weeks) or patients may also have spontaneous or iatrogenic preterm delivery. If the patient delivers before the 36th week or does not have data available in the 36th week, we will use the last available week of data If the patient does not have glucose log in the 36th week, we will use the most proximal week such as the 37th week.

SECONDARY OUTCOMES:
Birth weight in grams | At birth
  continuous measure birthweight in grams of neonate of the pregnancy as recorded in the delivery record
Fasting blood glucose >50% at target within the past week | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  categorical measure of fasting BG at target. Fasting blood glucose at target (>95) in greater than 50% of recorded values with in the past week
Postprandial blood glucose >50% at target within the past week | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  categorical measure of fasting BG at target. Postprandial blood glucose >50% at target (<140 at 1 hour postprandial or <120 at 2 hour postprandial) within the past week
Average fasting blood glucose | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  Continuous measure of average fasting blood glucose. Average fasting blood glucose for each week of the pregnancy from randomization until delivery
Average postprandial blood glucose | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  Continuous measure of average postprandial blood glucose. Average fasting blood glucose for each week of the pregnancy from randomization until delivery
Maternal hypoglycemia events | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  Number of maternal hypoglycemia events defined as percent fasting glucose below 60
Total insulin usage (units/kg/day) | at time of delivery approximately from 36 weeks to 39 weeks gestation
  continuous measure total insulin usage at time of delivery
Composite perinatal outcomes (large for gestational age, neonatal hypoglycemia, NICU admission) | At birth
  categorical measure of the presence composite outcomes of large for gestational age, and neonatal hypoglycemia and NICU admissions of as a result of pregnancy.
Neonatal hypoglycemia | at birth until 24 hours birth
  categorical measure if neonatal hypoglycemia is present as defined as blood glucose <35 mg/dL requiring glucose treatment in the first 24 hours of birth
NICU admissions | Any NICU admission for 48 hours or greater duration up to 2-3 months
  categorical measure if neonate is admitted to the neonatal intensive care unit for any indication at birth or until discharge of neonate
Preterm birth <34 weeks for any indication | At birth
  categorical measure of the presence of delivery before 34 weeks either spontaneous or iatrogenic
Preterm birth <37 weeks for any indication | At birth
  categorical measure of the presence of delivery before 37 weeks either spontaneous or iatrogenic
Hypertensive disorder of pregnancy | From randomization to delivery, which is approximately from 36 weeks to 39 weeks gestation
  categorical measure of the presence of the diagnosis of hypertensive disorder of pregnancy including gestational hypertension, preeclampsia with and without severe features, and superimposed preeclampsia, eclampsia, and HELLP syndrome as defined by ACOG guidelines
Large for gestational age | At birth
  Categorical measure if neonate is large for gestational age as defined by 90th percentile for birthweight standardized by gestational age and sex
Demographics and logistic barriers survey | after the 36th week until delivery
  continuous measure of survey from the demographics and logistic barriers survey
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | after the 36th week until delivery
  continuous measure of survey information from Diabetes Treatment Satisfaction Questionnaire (DTSQ) assessing patients' satisfaction with their diabetes treatment
Diabetes Distress Screening (DDS) Scale | after the 36th week until delivery
  continuous measure of survey Diabetes Distress Screening (DDS) Scale assessing the severity of the distress with living with gestational diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Venkatesh, MD, PhD, Principal Investigator — Ohio State University; Xiao-Yu Wang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center OB/GYN Maternal and Fetal Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] McGovern AP, Hirwa KD, Wong AK, Holland CJE, Mayne I, Hashimi A, Thompson R, Creese V, Havill S, Sanders T, Blackman J, Vaidya B, Hattersley AT. Patient-led rapid titration of basal insulin in gestational diabetes is associated with improved glycaemic control and lower birthweight. Diabet Med. 2022 Oct;39(10):e14926. doi: 10.1111/dme.14926. Epub 2022 Aug 8. PMID 35900879
- [Background] Bradley C, Plowright R, Stewart J, Valentine J, Witthaus E. The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc) evaluated in insulin glargine trials shows greater responsiveness to improvements than the original DTSQ. Health Qual Life Outcomes. 2007 Oct 10;5:57. doi: 10.1186/1477-7525-5-57. PMID 17927832
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2022. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2022 Nov 1;45(11):2753-2786. doi: 10.2337/dci22-0034. PMID 36148880